CLINICAL TRIAL: NCT03728088
Title: Non-technical Attributes and Surgical Experience: a Cross-sectional Study Comparing Communication Styles and Attitudes in Surgical Staff, Trainees and Applicants
Brief Title: Cross-sectional Analysis of Non-technical Attributes and Surgical Experience in Surgical Staff, Trainees and Applicants.
Status: Enrolling by invitation | Type: Observational
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: B670201628799
Record Dates: First submitted 2018-10-23; First posted 2018-11-01 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Healthy Volunteers
Keywords: Non-technical attributes; Surgical training; Communication style; Risk aversion; Reaction to uncertainty; Self-assessment

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Surgical Candidates: Under- and postgraduate candidates applying for surgical training in general surgery, orthopedics, urology or plastic surgery at Ghent University Hospital.
  All candidates will complete the rating scales concerning non-technical attributes in the period prior to the surgical selections.
  Interventions: Other: Rating scales concerning non-technical attributes
- Surgical trainees: Surgical trainees active in general surgery, orthopaedics, urology or plastic surgery, at Ghent University Hospital or an affiliated non-academic training hospital.
  All trainees will be invited to participate in the study. Trainees who agree to participate will complete the rating scales concerning non-technical attributes.
  Interventions: Other: Rating scales concerning non-technical attributes
- Surgical staff: Surgical staff members active in general surgery, orthopaedics, urology or plastic surgery, at Ghent University Hospital.
  All surgical staff members will be invited to participate in the study. Surgical staff members who agree to participate will complete the rating scales concerning non-technical attributes.
  Interventions: Other: Rating scales concerning non-technical attributes

INTERVENTIONS:
Other: Rating scales concerning non-technical attributes
  Other Names: Communication styles inventory (CSI-96) rating scale; Physician's reactions towards uncertainty (PRU) rating scale; Physicians's risk attitudes (PRA) rating scale

SUMMARY:
This study consists of an analysis of the communication styles and attitudes towards risk and uncertainty (i.e. non-technical attributes) in a surgical population with varying clinical experience.

The study aims to investigate the differences and specific patterns in non-technical attributes that may be discerned in these groups and how these non technical attributes develop throughout surgical training.

DETAILED DESCRIPTION:
This study evaluated the communication styles and attitudes towards risk and uncertainty in a population of surgical candidates (pre- and postgraduates), surgical trainees and surgical staff members, from the specialties of general surgery, orthopedics, urology and plastic surgery. After signing informed consent, participants complete an on-line questionnaire, which contains a set of validated tools.

Initially, a cross-sectional analysis of the non-technical attributes will be conducted, to identify any patters, similarities or differences between participant groups.

The study hypothesis is that significant differences can be observed in participant attributes, which relate to their clinical experience.

Additionally, surgical candidates who agree to participate in this study and are accepted for a surgical training in either general surgery, orthopaedics, urology or plastic surgery, will be invited to repeat the questionnaire at a 2-year interval, to investigate the evolution of their non-technical attributes throughout their training and to identify general patterns.

ELIGIBILITY:
Inclusion Criteria:

* Participant is part of any of the following groups:

  * Applicant for surgical training in general surgery, orthopedics, urology or plastic surgery.
  * Trainee in general surgery, orthopedics, urology, plastic surgery.
  * Staff in general surgery, orthopedics, urology, plastic surgery.
* Participant is active at Ghent University Hospital or an affiliated training hospital.

No exclusion criteria apply to this study.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Candidates applying for a surgical specialty (general surgery, orthopaedics, urology, plastic surgery); trainees in one of these surgical specialties; staff members in one of these surgical specialties.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2016-09-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Participant communication styles | Rating scale is completed by all groups on study inclusion, after signing informed consent.
  Communication Styles Inventory-96 scale:Subdomains: Expressiveness (range: 1-5); Preciseness (range: 1-5); Verbal aggressiveness (range: 1-5); Questioningness (range: 1-5); Emotionality (range: 1-5); Impression manipulativeness (range: 1-5)
Participant attitudes towards uncertainty | Rating scale is completed by all groups on study inclusion, after signing informed consent. For the candidate group, this measure is repeated on a selection day during the surgical selection process, +- 1 - 2 months after study inclusion
  Physicians' Reactions to Uncertainty (PRU) scale: Anxiety due to uncertainty (Range: 5-30
  ); Concern about bad outcomes (3-18); Reluctance to disclose uncertainty to patients (Range: 5-30); Reluctance to disclose mistakes to physicians (Range 2-12)
Participant attitudes towards taking risks | Rating scale is completed by all groups on study inclusion, after signing informed consent. For the candidate group, this measure is repeated on a selection day during the surgical selection process, +- 1 - 2 months after study inclusion
  Physicians' risk attitude (PRA) Scale (Range: 2-12)

SECONDARY OUTCOMES:
Participant perceived actual health status | Rating scale is completed by all groups on study inclusion, after signing informed consent.
  Short Form-36 scale (Range: 10-50)

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Van Herzeele, MD, PhD, Principal Investigator — Vascular surgeon

IPD SHARING:
Plan to Share IPD: No
Research data will not be shared standard.